CLINICAL TRIAL: NCT03712800
Title: Efficacy of Rhythmical Massage in Comparison to Heart Rate Variability Biofeedback in Women With Primary Dysmenorrhea - a Randomized, Controlled Trial
Brief Title: Rhythmical Massage Compared With Heart Rate Variability Biofeedback in Women With Menstrual Pain (Dysmenorrhea)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ARCIM Institute Academic Research in Complementary and Integrative Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DYS_01
Record Dates: First submitted 2018-10-18; First posted 2018-10-19 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: Primary Dysmenorrhea
Keywords: Dysmenorrhea; Women Health; Rhythmical Massage; Anthroposophic Medicine; HRV Biofeedback
MeSH Terms: conditions — Dysmenorrhea

STUDY DESIGN:
Intervention Model Description: Participants are randomized to one of the three groups (rhythmical massage, HRV biofeedback or control). After the three-month intervention period, the controls receive rhythmical massage for ethical and compliance reasons. Assessments are taken before and after the intervention phase. Pain intensity is once more queried three months after the end of the intervention period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Rhythmical massage (Experimental): Participants who receive rhythmical massage for three months.
  Interventions: Other: Rhythmical massage
- HRV biofeedback (Experimental): Participants who perform HRV biofeedback for three months.
  Interventions: Behavioral: HRV biofeedback
- Control group (No Intervention): Participants who do not receive an intervention during the three-month intervention period but are advised to stay with their usual care during menstrual pain. For ethical and compliance reasons, these participants receive a series of rhythmical massage treatments after the initial three-month intervention/control period.

INTERVENTIONS:
Other: Rhythmical massage — Rhythmical Massage according to Dr Ita Wegman, derived from Swedish Massage in the 1920s. Applied for various indications in the context of Anthroposophic Medicine, aiming at a recovery of self-regulation and self-healing forces.
  Arms: Rhythmical massage
Behavioral: HRV biofeedback — One of various biofeedback types, HRV biofeedback gives a visual feedback of the participant's heart rate variability as an indicator for general health, physical and cognitive performance, self-regulation and a decreased risk of illness.
  Arms: HRV biofeedback

SUMMARY:
A study to explore whether rhythmical massage and heart rate variability biofeedback can help to reduce pain in women suffering from menstrual pain (dysmenorrhea).

DETAILED DESCRIPTION:
This is a three-arm randomized controlled trial to evaluate the efficacy of rhythmical massage and HRV biofeedback in women with primary dysmenorrhea compared to a control group. The main focus is on pain intensity during menstruation. Moreover, analgesics intake, SF-12 mental and physical scores and parameters of a 24h-HRV measurement are assessed before and after the three-month intervention.

ELIGIBILITY:
Inclusion Criteria:

* At least one year of primary dysmenorrhea (physician-confirmed).
* Written informed consent (also from parents/legal guardians of underage girls).
* Menarche at least one year ago.

Exclusion Criteria:

* Secondary dysmenorrhea.
* Participation in another study.
* Mental retardation.
* Addiction.

Ages: 16 Years to 46 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Mean pain intensity during menstruation | Baseline (pre intervention) and after three months (post intervention).
  Mean pain intensity on the three days of maximal menstrual discomfort, as indicated by the participants on a numeric rating scale in a pain diary.

SECONDARY OUTCOMES:
Maximum pain intensity during menstruation | Baseline (pre intervention) and after three months (post intervention).
  Maximum pain intensity on the three days of maximal menstrual discomfort, as indicated by the participants on a numeric rating scale in a pain diary.
SF-12 sum-score | Baseline (pre intervention) and after three months (post intervention).
  Overall quality of life as assessed by the SF-12 questionnaire.
SF-12 mental | Baseline (pre intervention) and after three months (post intervention).
  Quality of life (subscore mental) as assessed by the SF-12 questionnaire.
SF-12 physical | Baseline (pre intervention) and after three months (post intervention).
  Quality of life (subscore physical) as assessed by the SF-12 questionnaire.
SDNN | Baseline (pre intervention) and after three months (post intervention).
  Standard deviation of normal to normal beats, derived from 24h ECGs.
RMSSD | Baseline (pre intervention) and after three months (post intervention).
  Root mean square of successive differences, derived from 24h ECGs.
LF/HF-Ratio | Baseline (pre intervention) and after three months (post intervention).
  LF/HF-Ratio = Ratio of two bands from frequency domain analysis: LF band (0.04-0.15 Hz), HF band (0.15-0.40 Hz), derived from 24h ECGs.
Analgesics intake during menstruation | Baseline (pre intervention) and after three months (post intervention).
  Percentage of participants taking analgesics.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Vagedes, MD, Dr, Principal Investigator — Arcim Institute
Locations (1):
- Die Filderklinik, Filderstadt, Baden-Wurttemberg, Germany